CLINICAL TRIAL: NCT02266784
Title: Smoking/Nicotine Dependence in Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Contingency Management, Quitting Smoking, and ADHD
Acronym: ADQUIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00055228; 2K24DA023464-06A1 (NIH)
Record Dates: First submitted 2014-10-09; First posted 2014-10-17 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cigarette Smoking; Smoking Cessation
Keywords: smoking, smoking cessation, contingency management, ADHD
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation; Smoking; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management (CM) (Experimental): ADHD (N=20) & CTRL (N=20). Participants will earn compensation, based upon smoking abstinence via a Contingency Management (CM) system. This level of compensation will increase by the same amount each visit based upon abstinence. In addition, escalating bonus payments will be available for evidence of continued abstinence. The first 10 visits will be daily weekdays. The following 9 visits will be over three weeks. The final 3 treatment visits will occur weekly. The 2nd & 3rd type visits CM payments will be based upon monitoring participants' cotinine levels. A missed visit or elevated CO level will lead to 1) no CM payment for that day; 2) resetting the contingencies such that the next CO sample that is below the criterion will result in payment equal to the first day. If there is a lapse, participants' contingencies will be reinstated at their previous highest level post 3 abstinent days. Also follow-up visits at 3 and 6 months.
  Interventions: Behavioral: Contingency Management (CM)
- Treatment as Usual (Other): ADHD (N=20). Transdermal nicotine skin patches (i.e. Habitrol) will be used along with supportive counseling in the treatment as usual groups. Visit schedules will coincide with the visit schedules for the CM groups (daily visits for 1st 2 weeks, 3X weekly visits for weeks 3-5, 1x weekly visit for weeks 6-8). A standard regimen of nicotine replacement with which the study team has experience will be used: four weeks of 21 mg/d beginning on the QD, two weeks of 14 mg/d and two weeks of 7 mg/d. Also follow-up visits at 3 and 6 months.
  Interventions: Drug: Transdermal nicotine skin patches (i.e. Habitrol); Other: Supportive Counseling

INTERVENTIONS:
Behavioral: Contingency Management (CM)
  Arms: Contingency Management (CM)
Drug: Transdermal nicotine skin patches (i.e. Habitrol)
  Arms: Treatment as Usual
Other: Supportive Counseling
  Arms: Treatment as Usual

SUMMARY:
The overall goal of the study is to evaluate how motivation and readiness for change are influenced in the context of a smoking cessation attempt. A total of 60 adult (i.e. age 18-55) smokers (N=40 with ADHD; N=20 without ADHD) who are interested in quitting will be enrolled into a 3-arm trial allocated as follows. Twenty of the ADHD smokers and the 20 non-ADHD smokers will be assigned to a traditional 8-week contingency management intervention in which monetary payments will be made contingent upon biologically verified evidence of smoking abstinence. The 20 additional ADHD smokers will be assigned to a treatment-as-usual condition (nicotine replacement; supportive counseling). During the treatment phase, subjects will be required to answer questions 4x/week in their daily lives via an EMA (Ecological Momentary Assessment).

Specific Aim 1: To assess motivation to quit smoking and readiness for change prior to a quit attempt in treatment seeking ADHD and non-ADHD smokers. Hypothesis 1a: The investigators hypothesize that prior to a quit attempt, smokers with ADHD will exhibit significantly lower levels of intrinsic motivation to quit, and equal or higher levels of extrinsic motivation to quit compared to smokers without ADHD. Hypothesis 1b: The investigators hypothesize that smokers with ADHD will exhibit relatively less readiness for change than smokers without ADHD.

Specific Aim 2: To assess how baseline levels of motivation to quit and readiness for change are influenced during a quit attempt as a function of both ADHD status and treatment modality. Hypothesis 2a. The investigators hypothesize that the CM intervention will result in relatively greater change in extrinsic motivation to quit versus intrinsic motivation to quit, and that this effect will be more pronounced among ADHD smokers. Hypothesis 2b: The investigators hypothesize that overall motivation to quit (intrinsic and extrinsic) and readiness for change will be significantly influenced by the CM intervention versus treatment as usual among ADHD smokers.

Exploratory Aim 1: To assess the relative efficacy of a CM intervention versus treatment as usual in smokers with ADHD. The investigators hypothesize that CM will be more effective for promoting short-term (4-8 weeks) smoking abstinence, as well as for promoting longer-term (3-6 months) smoking cessation.

Exploratory Aim 2: To assess the associations among smoking withdrawal/craving, affect, ADHD symptoms, and motivation to quit/readiness for change. The investigators hypothesize that higher levels of motivation and readiness for change will be associated with lower levels of self-reported withdrawal, craving, and negative affect.

DETAILED DESCRIPTION:
Individuals with ADHD have altered reinforcement/motivational functioning that are likely related to risk for smoking and recalcitrance for quitting. The investigators lab has demonstrated that the abstinence-induced reinforcing effects of cigarette smoking are more pronounced in ADHD smokers. However, in spite of these increases and demonstrated differences in withdrawal severity, interventions that provide reinforcement contingent on abstinence appear to work well for smokers with ADHD. To date, no studies have explicitly investigated how motivational processes are associated with smoking cessation attempts in ADHD smokers. The proposed pilot research is therefore highly innovative since it will evaluate how these processes change and influence outcomes during two different kinds of smoking cessation interventions. The project will also provide important pilot data on potential differences between ADHD and non-ADHD smokers in the context of a contingency management (CM) trial, which will help guide the development of more refined and targeted cessation interventions for this high risk group of smokers.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Male or female; if female of child-bearing potential, must be using an acceptable form of contraception
* ADHD Diagnosis:
* For ADHD Groups: confirmed primary diagnosis, any subtype as determined by the clinician administered CAADID and clinical interview
* For Control Group: NO diagnosis of ADHD as determined by clinician administered CAADID and clinical interview
* ADHD Symptom Ratings:
* For ADHD Groups: T-Score > 65 on one of the DSM-IV relevant scales (Inattentive Symptoms, Hyperactive-Impulsive Symptoms, Total Symptoms or ADHD Index) on both the Self-Report and Observer versions of the CAARS
* For Control Group: T-Score < 60 on all of the DSM-IV relevant scales (Inattentive Symptoms, Hyperactive-Impulsive Symptoms, Total Symptoms or ADHD Index) on both the Self-Report and Observer versions of the CAARS
* Self-report smoking at least 10 cigarettes/day
* Provides an afternoon exhaled carbon monoxide reading of at least 10 ppm.
* Cognitive functioning > 80 as assessed by the KBIT-II

Exclusion Criteria:

* History of chronic/significant medical condition
* Use of any psychoactive medication in the past 12 months, other than FDA-approved medication for the ADHD group only
* Estimated IQ < 80 on Kaufmann Brief Intelligence Test, Second Edition
* Has a primary diagnosis of any other Axis I Disorder (determined by the Structured Diagnostic Interview for DSM; SCID) that is significantly impairing and would contraindicate participation in the present study
* Has a primary diagnosis of any Axis II Disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Change in motivation to quit smoking, as measured by the Readiness to Change Questionnaire | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Readiness to Change Questionnaire (RCQ) is a measure designed to assess attitudes toward quitting smoking.
Change in motivation to quit smoking, as measured by the Treatment Self-Regulation Questionnaire | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Treatment Self-Regulation Questionnaire measures autonomous motivation.
Change in motivation to quit smoking, as measured by the Perceived Competence Scale for Cessation | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Perceived Competence Scale for Cessation measures perceived competence to quit.
Change in motivation to quit smoking, as measured by the Reasons For Quitting questionnaire | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Reasons For Quitting questionnaire measures relative levels of intrinsic versus extrinsic motivation to quit smoking.
Change in readiness to change behavior, as measured by the Readiness to Change Questionnaire | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Readiness to Change Questionnaire (RCQ) is a measure designed to assess attitudes toward quitting smoking.
Change in readiness to change behavior, as measured by the Treatment Self-Regulation Questionnaire | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Treatment Self-Regulation Questionnaire measures autonomous motivation.
Change in readiness to change behavior, as measured by the Perceived Competence Scale for Cessation | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Perceived Competence Scale for Cessation measures perceived competence to quit.
Change in readiness to change behavior, as measured by the Reasons For Quitting questionnaire | Baseline to 9 weeks
  During the treatment period, participants will answer at least 4 times weekly, questionnaires to assess motivation for behavior change, autonomy, and interest in quitting. The Reasons For Quitting questionnaire measures relative levels of intrinsic versus extrinsic motivation to quit smoking.
Comparison of populations in motivation to quit on the Reasons for Quitting Questionnaire | Baseline to 9 weeks
  The study team will compare the change in scores for extrinsic and intrinsic motivation to quit on the Reasons for Quitting Questionnaire in the ADHD and non-ADHD groups assigned to receive CM.

SECONDARY OUTCOMES:
Change in smoking behavior in ADHD population | Baseline, 3 months, 6 months
  This outcome is based both upon the treatment period and follow-up visits at 3 and 6 months. CM is proposed to be a potential more effective treatment in an ADHD population in the short and longer term, in comparison to treatment as usual. This will be measured by urine cotinine level and residual Carbon Monoxides levels from samples provided by participants.
Decreasing effects of quitting smoking. | Baseline, 3 months, 6 months
  This outcome assesses overall whether increased motivation and readiness for behavior change (i.e. quit smoking), potentially associated CM, will decrease negative aspects of quitting. These include smoking withdrawal/craving, affect, and impact on ADHD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Kollins, Ph.D., Principal Investigator — Duke Health
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States